CLINICAL TRIAL: NCT05241054
Title: Comparison of Local Anesthesia and Induced Hypotensive Anesthesia on Quality of External Dacryocystorhinostomy Operation Under General Anesthesia
Brief Title: Effect of Local Anesthesia Versus Induced Hypotensive Anesthesia on Quality of External Dacryocystorhinostomy Operation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MD / 21.09.536
Record Dates: First submitted 2022-01-24; First posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-01

CONDITIONS: Patient With Nasolacrimal Duct Obstruction; External Dacryocystorhinostomy Operation
MeSH Terms: interventions — Bupivacaine; Nitroglycerin; Propofol; Fentanyl; Atracurium; Respiration, Artificial; Sevoflurane; Ringer's Lactate; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double-blind study (patient and data collector)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bupivacaine (Active Comparator): Patients will receive local anesthesia by paranasal infiltration at the incision site with 2.5 ml of 0.5% bupivacaine with 1:100000 epinephrine.
  Interventions: Drug: Bupivacaine; Drug: Propofol; Drug: Fentanyl; Drug: Atracurium Besylate; Procedure: Mechanical ventilation; Drug: Sevoflurane; Drug: Lactated Ringers; Other: Head-up tilt; Drug: Paracetamol
- Nitroglycerine (Active Comparator): Patients will receive an infusion of Nitroglycerine (TNG) (0.2-1μg/kg/min) will be started and adjusted to maintain mean arterial blood pressure between 55-65 mmHg.
  Interventions: Drug: Nitroglycerine; Drug: Propofol; Drug: Fentanyl; Drug: Atracurium Besylate; Procedure: Mechanical ventilation; Drug: Sevoflurane; Drug: Lactated Ringers; Other: Head-up tilt; Drug: Paracetamol

INTERVENTIONS:
Drug: Bupivacaine — With patient in supine position, the patient will be placed on the operating table with a head-up tilt to reduce venous congestion at the operative site. Skin will be disinfected, the patient will receive local anesthesia by paranasal infiltration at the incision site with 2.5 ml of 0.5% bupivacaine with 1:100000 epinephrine.
  Arms: Bupivacaine
Drug: Nitroglycerine — This group includes 32 patients (anticipated), infusion of Nitroglycerine (TNG) (0.2-1µg/kg/min) will be started and adjusted to maintain mean arterial blood pressure between 55-65mmHg.
  Arms: Nitroglycerine
Drug: Propofol — General anesthesia will be induced using IV propofol at dose of 1-2 mg.kg
Drug: Fentanyl — fentanyl 1 microgram.kg
Drug: Atracurium Besylate — Atracurium besylate 0.5mg.kg to facilitate intubation followed will top up dose of atracurium(0.1mg/kg).
Procedure: Mechanical ventilation — Patient will then be mechanically ventilated using a volume control mode with tidal volume 6-8ml/kg, respiratory rate 10-14 breath/min and I.E ratio1:2 to maintain end tidal CO2 around 35 mmHg
Drug: Sevoflurane — Anesthesia will then be maintained using sevoflurane 2%, and 60% air in oxygen mixture and top up dose of
Drug: Lactated Ringers — Intravenous infusion of Lactated Ringers will be given per body weight and according to intraoperative loss
Other: Head-up tilt — The patient is placed on the operating table with a head-up tilt to reduce venous congestion at the operative site
Drug: Paracetamol — paracetamol infusion (15 mg/kg) will be given by IV infusion in both groups

SUMMARY:
Bleeding is one of the important complications during Dacryocystorhinostomy, which dissatisfy ophthalmic surgeon, reduces surgical field visualization, and increases the duration of surgery Thus, the management of this complication is a great consideration during this operation. The aim of this study is to compare the efficacy of combined local and general anesthesia in a group of patients undergoing external dacryocystorhinostomy (DCR) operation versus the efficacy of general anesthesia with induced hypotensive anesthesia

DETAILED DESCRIPTION:
Dacryocystorhinostomy or DCR is among the common oculoplastics surgeries performed for managing epiphora due to nasolacrimal duct obstruction. The main purpose of DCR surgery is to eliminate the obstruction and to accomplish normal tear. DCR is a procedure performed to drain the lacrimal sac in which lacrimal flow is diverted into the nasal cavity through an artificial opening made at the level of the lacrimal sac in cases of chronic dacryocystitis or symptomatic nasolacrimal duct obstruction not relieved by simple probing and stringing.

Dacryocystorhinostomy (DCR) operation can be performed externally or endoscopically. External DCR was first described by Toti and this procedure was modified with the use of flaps by many authors. It is the gold standard of treatment with a reported success rate of more than 90%.

Bleeding during dacryocystorhinostomy (DCR) is trivial, but because of the anatomical vessel variation and presence of tiny vessels in the field of DCR, it can obscure the surgical field and complicate the operation.

One of the effective approaches for controlling bleeding tendency during DCR is to reduce blood pressure in patients. Ideal hypotensive medications administered to reduce blood pressure should have specific features such as easy to administration, being with rapid onset and offset without side effects, rapid elimination without any toxic metabolites, and having a predictable and dose-dependent action. Nitroglycerine (TNG) is a direct vasodilator agent, especially in veins, and produces hypotension, and is preferred by clinicians because of rapid onset and offset time and easy titration.

Another mechanism for controlling bleeding is infiltrating the incision site by local anesthetic with admixed epinephrine to promote local vasoconstriction to decrease blood loss and prolong the duration of local anesthesia providing more time for analgesia.

In this study, the investigators will compare the efficacy of local versus induced hypotensive anesthesia in generally anesthetized patients undergoing external DCR operation on amount of blood loss, quality of the surgical field, intraoperative hemodynamics, and surgeon satisfaction

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I and II
* patients who are scheduled for external Dacryocystorhinostomy operation

Exclusion Criteria:

* Patient refusal.
* Patients with history for cerebrovascular.
* Patients with history for coronary insufficiency.
* Local skin infection at site of injection.
* Known hypersensitivity to the study drugs.
* Extremes of age.
* Patients with any type of arrhythmias.
* Hematological diseases.
* Bleeding abnormality
* Coagulation abnormality

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Average category scale (ACS) | after 10 min of maintaining mean arterial blood pressure (MAP) at the desired range (55-65 mmHg)
  Assessment of intraoperative blood loss and quality of surgical field by Average category scale (ACS) for assessment of intraoperative surgical field (0-5): 0 - No bleeding 1 - Slight bleeding - no suctioning of blood required 2 - Slight bleeding 3- slight bleeding required suctioning 4- moderate bleeding 5- sever bleeding

SECONDARY OUTCOMES:
Mean arterial blood pressure | procedure (basal reading and every 5 minutes till the end of anesthesia )
  Mean arterial blood pressure values will be recorded
Heart Rate (HR) | procedure (basal reading and every 5 minutes till the end of anesthesia)
  Heart Rat values will be recorded
Postoperative visual analogue score (VAS) | up to 24 hours after the procedure
  Pain levels will be assessed post operatively using visual analogue score (vas) at 0 min , 6 hour, 12hour , 24hours postoperatively .
Postoperative analgesics intake | up to 24 hours after the procedure
  Total dose of ketorolac requirements will be recorded
Surgeon satisfaction | at the end of the procedure
  Surgeon satisfaction will be recorded based on a 4 points scale (1=bad, 2=moderate, 3=good, 4=excellent).
Nausea | up to 24 hours after the procedure
  Postoperative Nausea will be assessed on a scale of 0 to 3 [0; no nausea, 1, mild nausea, 2; moderate nausea, 3; severa nausea]
Vomiting | up to 24 hours after the procedure
  Postoperative Vomiting will be assessed on a scale of 0 to 3 [0; no vomiting, 1, mild vomiting, 2; moderate vomiting, 3; severe vomiting]
Hematoma | up to 24 hours after the procedure
  The patients will be evaluated postoperatively to identify the occurrence of hematoma (blood collection, swelling, bruises) at the site of injection of bupivacaine.

CONTACTS AND LOCATIONS:
Overall Officials: Ola T Abdel Dayem, MD, Study Chair — Professor, MD anesthesia Department, Faculty of Medicine, Mansoura University, Egypt; Hazem Moawad, MD, Study Director — Assistant professor, MD anesthesia Department, Faculty of Medicine, Mansoura University, Egypt
Locations (1):
- Mansoura University, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The individual data sharing strategy. The data that support the findings of this study will be available on request from a principal investigator
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After six months after completing the study.